CLINICAL TRIAL: NCT07398521
Title: A Clinical Trial to Evaluate the Effects of a Supplement on Energy and Mood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cymbiotika, LLC (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20811
Record Dates: First submitted 2026-02-04; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Mood; Stress
Keywords: Sleep Quality; Magnesium
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liposomal Magnesium Complex (Experimental): Participants will consume one packet daily by squeezing the contents directly into the mouth.
  Interventions: Dietary Supplement: Liposomal Magnesium Complex

INTERVENTIONS:
Dietary Supplement: Liposomal Magnesium Complex — The supplement is taken in the morning with the first meal of the day for 14 consecutive days.

SUMMARY:
This study evaluates the effects of a Liposomal Magnesium Complex supplement on energy and mood. The study is a single-arm, virtual trial in which 60 adult participants consume the supplement daily for 14 days and complete self-reported questionnaires at multiple timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female
* Be aged 18-60
* Anyone currently experiencing issues regarding all of the following: Low energy, Difficulty regulating mood
* Anyone who is generally healthy - does not live with any uncontrolled chronic disease.
* Anyone willing to avoid all other dietary supplements or products containing magnesium for the duration of the trial.
* Anyone willing to refrain from taking any products, prescription medications, or supplements that target energy, mood, stress, and sleep during the test period.
* Anyone willing to maintain their current diet, sleep schedule, and activity level for the duration of the study.
* Resides in the United States.

Exclusion Criteria:

* Anyone with pre-existing chronic conditions that would prevent participants from adhering to the protocol, including cancer and mental health disorders.
* Anyone with a nut allergy or allergies or sensitivities to any of the product ingredients.
* Any women who are pregnant, breastfeeding, or trying to conceive (or who will be at any point during the study period).
* Anyone who drinks heavily (i.e., 8 or more alcoholic drinks per week for women or 15 or more alcoholic drinks per week for men).
* History of diagnosed psychiatric or mood disorders.
* History of diagnosed sleep disorders.
* History of serious illness in the last three months.
* History of substance abuse.
* History of kidney disease.
* History of hormone or endocrine disorders, including but not limited to hypothyroidism, Hashimoto's thyroiditis, polycystic ovarian syndrome (PCOS), and diabetes.
* Planned surgery during the study period.
* Currently partaking in another research study or will be partaking in any other research study for the next 2 weeks, or at any point during this study's duration.
* Anyone unwilling to follow the study protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-10-14 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Change in Energy Levels | Baseline, Day 3, Day 7, Day 10, Day 14
  Change in self-reported energy levels following daily use of the Liposomal Magnesium Complex supplement, assessed using participant questionnaires.
Change in Mood | Baseline, Day 3, Day 7, Day 10, Day 14
  Change in self-reported mood following daily use of the Liposomal Magnesium Complex supplement, assessed using participant questionnaires.

SECONDARY OUTCOMES:
Change in Stress Levels | Baseline, Day 3, Day 7, Day 10, Day 14
  Participant-reported changes in perceived stress levels assessed via questionnaire.
Change in Relaxation and Calmness | Baseline, Day 3, Day 7, Day 10, Day 14
  Participant-reported changes in feelings of relaxation and calmness assessed via questionnaire.
Change in Balanced Mood | Baseline, Day 3, Day 7, Day 10, Day 14
  Participant perception of mood balance assessed using self-reported questionnaires.
Change in Sleep Quality | Baseline, Day 3, Day 7, Day 10, Day 14
  Participant-reported changes in sleep assessed via questionnaire.
Change in Muscle Tension | Baseline, Day 3, Day 7, Day 10, Day 14
  Participant-reported changes in muscle tension assessed using questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No